CLINICAL TRIAL: NCT03665077
Title: Pilot Trial to Evaluate Blood and Imaging Based Biomarkers for Aromatase Inhibitor Induced Musculoskeletal Syndrome
Brief Title: Evaluation of Blood/Imaging Based Biomarkers, Aromatase Inhibitor Induced Musculoskeletal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1712078374; NCI-2018-00099 (Registry Identifier: NCI Trial Identifier)
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Aromatase Inhibitor Induced Musculoskeletal Syndrome (AIMSS); Breast Cancer
Keywords: Aromatase Inhibitor Induced Musculoskeletal Syndrome; AIMSS; Breast Cancer; Biomarkers; Oxylipin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants (Experimental): Patients with breast cancer who have completed all their primary treatments (surgery±radiation therapy) and are scheduled to start their adjuvant hormonal therapy.
  Interventions: Diagnostic Test: Initial blood draw; Diagnostic Test: Initial SWE ultrasound; Diagnostic Test: Blood draw at three months; Diagnostic Test: Blood draw at six months; Diagnostic Test: SWE ultrasound at six months

INTERVENTIONS:
Diagnostic Test: Initial blood draw — At baseline, patients will undergo a blood draw.
Diagnostic Test: Initial SWE ultrasound — At baseline, patients will undergo a sheer wave elastrography (SWE) ultrasound of their hands including wrists.
Diagnostic Test: Blood draw at three months — Blood drawn at three months to evaluate oxylipins.
Diagnostic Test: Blood draw at six months — Blood drawn at six months to evaluate oxylipins.
Diagnostic Test: SWE ultrasound at six months — SWE ultrasound at six months to evaluate tendon stiffness.

SUMMARY:
This is a pilot trial to evaluate for blood and imaging biomarkers in patients with breast cancer scheduled to start adjuvant hormonal therapy.

DETAILED DESCRIPTION:
This is a prospective single arm study enrolling patients (n = 25) with breast cancer scheduled to start adjuvant hormonal therapy. Patients would have completed all their primary treatments (surgery± radiation therapy) and are scheduled to start their adjuvant hormonal therapy. They get baseline blood drawn for oxylipins and sheer wave elastrography (SWE) ultrasound of their hands including wrists. They start adjuvant anastrozole and have blood drawn at 3mths and 6mths for measurement of oxylipins. SWE ultrasound is repeated at 6mths. This is a pilot trial to evaluate for blood and imaging biomarkers. Once pilot data is analyzed, goal is to apply for funding for a larger trial to further evaluate and validate these biomarkers

ELIGIBILITY:
Inclusion Criteria:

1. Be capable of understanding the investigational nature of the study and all pertinent aspects of the study
2. Be capable of signing and providing written consent in accordance with institutional and federal guidelines
3. Have a histologically-confirmed diagnosis of breast cancer
4. Be willing and able to comply with scheduled visits, treatment plan, and SWE ultrasound imaging
5. Age ≥ 21 years
6. Post-menopausal women with 1st event of ER+ early stage breast cancer (0-3)
7. Completed definitive therapy (surgery ± radiation)
8. Candidates for adjuvant AI therapy

Exclusion Criteria:

1. Have received adjuvant or neo-adjuvant chemotherapy
2. Prior endocrine therapy (AI or tamoxifen)
3. History of rheumatoid arthritis or other autoimmune arthritis
4. Daily non-steroidal anti-inflammatory drug (NSAID) use (except for daily aspirin use)
5. Current use of daily corticosteroids or immunosuppressive therapies

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Post-menopausal women
Enrollment: 28 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Oxylipins as Biomarkers for Aromatase Inhibitor-Induced Arthralgia (AIA) in Breast Cancer Patients — https://pubmed.ncbi.nlm.nih.gov/36984892/
- See also: Feasibility Trial to Evaluate Tendon Stiffness Obtained from Shear Wave Elastography Imaging as a Biomarker of Aromatase Inhibitor-Induced Arthralgias — https://pubmed.ncbi.nlm.nih.gov/35207339/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women with early-stage breast cancer prior to starting adjuvant endocrine therapy with aromatase inhibitors
Pre-assignment Details: This is a single arm observational study
Period: Overall Study
Arm/Group | Participants
Started | 28
3 Months Blood Draw | 22
6 Months Blood Draw | 24
Completed | 24
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 15
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 66.0 [63.1 to 72.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 28
Stage of Cancer [Count of Participants; unit: Participants] — Staging is based on the patients' surgical pathology report. American Joint Committee on Cancer (AJCC) 7th staging criteria for breast cancer was used for this study. Overall 7th Edition AJCC stage (IIV) is based on the TNM classification. The lower the number, the lower the cancer stage and the better the prognosis for the patient. The higher the stage, the worse the prognosis.
  Participants
    Stage 0 | 8
    Stage 1 | 17
    Stage 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Oxylipin Levels
Description: Change Oxylipin levels at Baseline, Three and Six Months
Time Frame: Baseline, Three months, and Six months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Participants
Number analyzed (Participants) | 24
pg/mL
  Baseline | 10.2 (5.9)
  3 Months | 12.1 (7.8)
  6 Months | 12.3 (9.8)
Statistical Analysis 1: Comparison: Participants; Test type: Other — Linear mixed-effect model of log-transformed oxylipin level, with time (date) as a continuous variable, adjusted for batch and clustered on participant; p = 0.684, Mixed Models Analysis; Linear mixed-effect model of log-transformed oxylipin level: time (date) as a continuous variable, adjusted for batch and clustered on participant

2. Secondary Outcome: Tendon Stiffness
Description: Tendon stiffness at baseline
Time Frame: Baseline
Population: Patients with breast cancer on adjuvant aromatase inhibitor.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Participants
Number analyzed (Participants) | 16
m/s
  Abductor pollicis longus (Baseline) | 5.59 (2.46)
  Median nerve (Baseline) | 5.56 (2.08)
Statistical Analysis 1: Comparison: Participants; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.02, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Pain Levels
Description: Pain levels at baseline and 6 months. Pain assessment was done using the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index; the WOMAC pain assessment consists of 5 items, and each item has a scale that ranges from 0-4 (higher scores indicate higher pain levels). The scores of the 5 items are summed up to obtain the WOMAC-total pain score, which ranges from 0-20.
Time Frame: Baseline, Six months
Population: Patients with early stage breast cancer on adjuvant aromatase inhibitor.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants
Number analyzed (Participants) | 24
score on a scale
  Baseline | 8.0 (14.6)
  6 Months | 12.3 (17.6)
Statistical Analysis 1: Comparison: Participants; Test type: Other — Linear mixed-effect model of log-transformed oxylipin level: time (date) as a continuous variable, adjusted for batch and clustered on participant; p = 0.058, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months.
Description: This is a pilot trial to evaluate oxylipins as blood biomarkers of aromatase inhibitor induced musculoskeletal syndrome. Adverse events were monitored for blood draws and analysis of oxylipins only. Anastrozole treatment was done as standard of care, and thus, side effects from anastrozole were managed per patients' standard of care and were not recorded for the purposes of this study.
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT03665077/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT03665077/ICF_001.pdf